CLINICAL TRIAL: NCT05328180
Title: aDjunct bicarbonatE in Local anaesthesIa for CarpAl Tunnel rElease (DELICATE): A Randomized Controlled Trial
Brief Title: aDjunct bicarbonatE in Local anaesthesIa for CarpAl Tunnel rElease (DELICATE)
Acronym: DELICATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5203139
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Release; Bicarbonate; Local anaesthesia; Wide awake lidocain cum adrenalin no tourniquet; Pain; Carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: Two concurrent study groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study nurse prepares the anaesthetic solution in advance, without reporting the contents to the surgeon or assisting nurses. The solution is labelled so that the surgeon doesn't know which solution is used. The used solution is recorded on a data pool and revealed only after the data analysis is made. Neither the investigators or outcome assessors have access to the randomized treatment before data has been analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-buffered local anaesthetic (Other): The investigators allocate 58 patients in this arm. It serves as the control group, who receives currently used local anaesthetic solution.
  Interventions: Other: Control arm
- Buffered local anaesthetic (Experimental): The investigators allocate 58 patients in this arm. It serves as the experimental group, who receives currently used anaesthetic solution that has been buffered.
  Interventions: Other: Sodium bicarbonate

INTERVENTIONS:
Other: Sodium bicarbonate — A 50/50 solution of lidocaine with adrenalin 1% and bupivacaine with adrenalin 0.5% is buffered with 7.5% sodium bicarbonate in 1:10.
  Arms: Buffered local anaesthetic
Other: Control arm — A 50/50 solution of lidocaine with adrenalin 1% and bupivacaine with adrenalin 0.5%.
  Arms: Non-buffered local anaesthetic

SUMMARY:
Introduction Carpal tunnel syndrome (CTS) is the most common peripheral nerve entrapment syndrome in Finland and worldwide. Nowadays carpal tunnel release (CTR) surgery is often done in local anaesthesia. Often the most painful event during CTR is the injection of the local anaesthetic. Multiple different methods have been trialed and buffering the local anaesthetic seems to have good results in reducing the pain caused by the injection. However, no study has buffered long-acting local anaesthetic in CTR surgery, and no study has accounted for the patient's individual pain tolerance in the groups. There are no comparisons of the results to minimal clinically important difference (MCID) for pain.

Hypothesis In this study the investigators will evaluate the effects of buffering long-lasting local anaesthetic in wide-awake local anaesthesia no tourniquet (WALANT) CTR. This study's hypothesis is that buffering long-acting local anaesthetic with sodium bicarbonate decreases the pain of the injection.

The investigators also expect that buffering will reduce the number of needle stings felt during injection, will result in as good perioperative pain control, will lengthen the effect of anaesthetic, will reduce postoperative painkiller usage, will have at least as good functional outcome and greater patient satisfaction.

Methods This study will enlist 116 patients and divide the patients into two groups in this double blinded randomized controlled trial. One group receives non-buffered, and the second group buffered local anaesthetic. This study's primary outcome is to compare burning, pressure, needle sting and total pain the patient experienced between the groups. The investigators will assess this using VAS, and will compare the results to MCID. The investigators secondary outcomes are comparisons of expected injection pain level and pain during CTR with VAS, individual pain tolerance/catastrophising tendency with preoperative PCS-FINv2.0 form, the number of needle stings the patient feels during the injection, functional outcome and improvement of the patients' symptoms with The Boston Carpal Tunnel Questionnaire (Likert 5) before and after the surgery, evaluation of patient satisfaction with net promoter score (NPS) and the use of painkillers, duration of analgesia and pain levels using VAS after the surgery until the 3rd postoperative night.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and electrophysiologically diagnosed carpal tunnel syndrome
* Patients who are scheduled for carpal tunnel release surgery.

Exclusion Criteria:

* Associated disease or conditions, including earlier injury to median nerve, cervical radiculopathy, cubital tunnel syndrome and other peripheral neuropathy
* Chronic renal failure
* Rheumatoid arthritis
* Allergies to lidocaine
* Pregnancy
* Profound cognitive impairment
* Previous ipsilateral carpal tunnel decompression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total pain level with visual analogic scale (VAS) | VAS is recorded immediately after the injection of local anaesthetic.
  The investigators evaluate the total pain with 0-100 mm visual analogue scale (VAS). In VAS higher number means more pain and is therefore worse. The investigators calculate the mean VAS level for each group and compare the results to find statistically and clinically relevant difference. Clinically relevant difference is evaluated by comparing the VAS difference to MCID.

SECONDARY OUTCOMES:
Burning pain level with VAS | VAS is recorded immediately after the injection of local anaesthetic.
  The investigators evaluate the total pain with 0-100 mm visual analogue scale (VAS). In VAS higher number means more pain and is therefore worse.
Pressure pain level with VAS | VAS is recorded immediately after the injection of local anaesthetic.
  The investigators evaluate the total pain with 0-100 mm visual analogue scale (VAS). In VAS higher number means more pain and is therefore worse.
Needle sting pain level with VAS | VAS is recorded immediately after the injection of local anaesthetic.
  The investigators evaluate the total pain with 0-100 mm visual analogue scale (VAS). In VAS higher number means more pain and is therefore worse.
CTR pain level | VAS is recorded right after CTR surgery
  The investigators evaluate the maximum pain level patient experiences during CTR surgery with visual analogue scale (VAS). This study uses 0-100 mm VAS. In VAS higher number means more pain and is therefore worse.
Analgesia duration | Every 4 hours after the surgery until 3rd postoperative night.
  The investigators assess the length of the anaesthesia by recording the pain level with visual analogue scale (VAS) every 4 hours. This study uses 0-100 mm VAS. In VAS higher number means more pain and is therefore worse.
Painkiller consumption | After the surgery until 3rd postoperative night.
  The investigators record the painkiller consumption after the surgery.
Number of needle stings | Immediately after the injection of local anaesthetic.
  The investigators ask the patient to report how many needle stings the patient felt during the injection of the local anaesthetic.
Pain catastrophizing tendency | Before the surgery.
  The investigators ask the patients to fill pain catastrophizing tendency evaluating form (PCS-FINv2.0) before the surgery in order to evaluate the pain levels between the experimental and control group. It has 13 questions and scores between 0-52. Higher score means higher pain catastrophizing tendency.
Functional outcome | Before and 3 months after the surgery.
  The investigators ask the patients to evaluate symptoms and functional outcome using the Boston Carpal Tunnel Questionnaire (BTCQ). It has 11 questions for symptoms of carpal tunnel syndrome and scores between 11 and 55. Higher score means more symptoms. BTCQ also has 8 questions for functionality of hand and it has scores between 8 and 40. Higher scores mean worse function of the hand.
Patient satisfaction | 3 months after the surgery.
  The investigators ask the patients to evaluate the surgery experience with net promoter score (NPS). NPS has 10 steps and higher value indicates greater satisfaction.
Expected pain level | Before the surgery.
  The investigators ask the patients to evaluate the pain the patient expect to experience during administration of local anaesthetic using visual analogue scale (VAS). This study uses 0-100 mm VAS. In VAS higher number means more pain and is therefore worse.

CONTACTS AND LOCATIONS:
Overall Officials: Yrjänä Nietosvaara, Prof., Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University hospital, Department of Orthopaedics, Traumatology and Hand Surgery, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
The investigators share pseudonymised data in EU/ETA if it is separately requested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 15 years after the study has ended.
Access Criteria: Request must come from an EU/ETA country. The investigators do not share data outside these countries.

REFERENCES:
- [Derived] Hytonen M, Nietosvaara Y, Reito A, Sirola J, Heikkinen N, Savolainen A, Raisanen MP. Protocol for a double-blinded randomised controlled trial investigating the use of adjunct bicarbonate in carpal tunnel release: a single-centre study. BMJ Open. 2023 Sep 18;13(9):e071488. doi: 10.1136/bmjopen-2022-071488. PMID 37723109

DOCUMENTS (1):
  • Informed Consent Form (2024-01-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT05328180/ICF_001.pdf